CLINICAL TRIAL: NCT05300542
Title: Efficacy Study of a Novel Cosmetic Product to Reduce an UVB Induced Erythema
Brief Title: Efficacy Study of a Novel Skin Health Product to Reduce an UVB Induced Erythema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 22.02.AMZ; 22.0103-65 (Other: proderm)
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Erythema; Sun Damaged Skin; Skin Inflammation
MeSH Terms: conditions — Erythema; Dermatitis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skin UVB irradiated 1.25MED (Experimental)
  Interventions: Other: Topical Placebo Cream; Other: Topical Cream with 0.5% Active; Other: Topical Cream with 1% Active
- Skin UVB irradiated 1.6MED (Experimental)
  Interventions: Other: Topical Placebo Cream; Other: Topical Cream with 0.5% Active; Other: Topical Cream with 1% Active
- Untreated Skin (No Intervention)

INTERVENTIONS:
Other: Topical Placebo Cream — Application of test products before and after irradiation
  Arms: Skin UVB irradiated 1.25MED; Skin UVB irradiated 1.6MED
Other: Topical Cream with 0.5% Active — Application of test products before and after irradiation
  Arms: Skin UVB irradiated 1.25MED; Skin UVB irradiated 1.6MED
Other: Topical Cream with 1% Active — Application of test products before and after irradiation
  Arms: Skin UVB irradiated 1.25MED; Skin UVB irradiated 1.6MED

SUMMARY:
The aim of this study is to determine the erythema-reducing efficacy of a test product in two concentrations on a light sunburn induced by a sun simulator compared to an untreated control and a placebo product.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and/or male
* From 18 to 65 years of age
* Uniform skin color and no erythema or dark pigmentation in the test area
* ITA° > 28 in the test area

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Insulin-dependent diabetes mellitus
* Electronic implant (e.g. pace maker, insulin pump, hearing aid, and the like) that cannot be removed during irradiation
* Documented allergies to cosmetic products and/or ingredients
* Active skin disease at the test area
* Irregularly tanned skin in the test area
* Medical history of dysplastic nevi, melanoma or other skin carcinoma
* Medical history of abnormal response to sunlight
* Regular use of tanning beds (more than 10 times within the last 6 months)
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Usage of medication with known photo-toxic and/or photo-sensitizing potential (e.g. some antibiotics, blood pressure regulating agents and antidepressants agents; hypericum perforatum) within the last 14 days prior to the start of the study and/or throughout the entire course of the study
* Any topical medication at the test area within the last 7 days prior to the start of the study and/or throughout the entire course of the study
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) within the last 7 days prior to the start of the study and/or throughout the entire course of the study
* Systemic therapy with anti-phlogistic agents or analgetics (e.g. diclophenac), except for minor pain relief medicine like acetylsalicylic acid or paracetamol within the last 3 days prior to the start of the study and/or throughout the entire course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Erythema (skin redness) assessed by Chromameter | 3 days
Visual erythema evaluation by a trained grader on a scale of -2 (marked redness) to 3 (no redness) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Klaus-Peter Wilhelm, Dermatologist, MD, Study Chair — proDERM GmbH; Dr. rer. nat. Sabrina Laing, MD, Principal Investigator — proDERM GmbH
Locations (1):
- proderm GmbH, Schenefeld, Germany